CLINICAL TRIAL: NCT06979128
Title: PICC Inserted by a Nurse-led Vascular Access Team in Poland
Acronym: NIce-PICC
Status: Recruiting | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Other Study IDs: KB/35/2025
Record Dates: First submitted 2025-05-07; First posted 2025-05-18 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-05

CONDITIONS: Vascular Access; PICC Line Placement
Keywords: PICC; peripherally inserted central catheter; chest x-ray; PICC tip navigation; nurse; vascular access team
MeSH Terms: interventions — Catheterization, Peripheral

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who requrie a PICC: All subjects patients who requrie a PICC
  Interventions: Procedure: PICC placement

INTERVENTIONS:
Procedure: PICC placement — Patient scheduled for PICC placement

SUMMARY:
Implantation of PICCs by a trained, dedicated nursing team can be effective and safe, and allows for intravenous therapy that requires medium- to long-term central venous access.

DETAILED DESCRIPTION:
The insertion of Peripherally Inserted Central Catheters (PICCs) offers numerous advantages over direct puncture of central veins. Ultrasound-guided insertion of PICCs into the peripheral vein is characterized by the high efficiency and safety of the procedure as well as patient comfort, and is a safe alternative to centrally inserted central catheters (CICCs) associated with a lower risk of complications. The PICCs will be inserted into one of the veins of the arm (basilic, brachial, cephalic) under ultrasound guidance. Cannulation will be supervised by a physician. Prior to cannulation a local anesthetic drug will be applied to the site of the planned puncture. Each PICC cannulation set consists of an echogenic needle, a guidewire, an introducer, a catheter with a diameter of 4 or 5 Fr and a length of 50-60 cm, a adhesive sutureless fixation, a semi-permeable transparent dressing, a needleless connector and a sticker indicating the type of vascular access. During the procedure intracavitary ECG will be used to catheter tip navigation. After the procedure, a chest X-ray will be taken to document the correct position of the tip. Taking into account the experience of the researchers and the learning curve described in the literature, it is planned to perform 200 PICC insertion procedures during the study period (50 per operator).

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Intravenous therapy with solutions requiring central vein cannulation (irritant drugs, extreme pH <5 and >9, osmolarity > 600 mOsm/l), e.g., chemotherapy, parenteral nutrition with osmolarity >900 mOsm/l
* Difficult intravenous access with multiple blood collection
* Ability to consent to participate in the study
* Consent to participate in the study

Exclusion Criteria:

* Presence of central venous catheter, such as. centrally inserted central catheter or totally implanted vascular device
* Indication of another type of vascular access device
* Lack of veins suitable for cannulation of the arm
* Infection, burns or other skin lesion on the upper extremities (involving the site of planned catheter insertion and attachment)
* Pregnancy (confirmed by history and review of medical records or confirmed by positive human chorionic gonadotropin (hCG) determination in urine or plasma)
* Lack of patient consent to participate in the study
* Lack of capacity to consent to participate in the study
* No physician present to supervise the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects patients who require a PICC
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
First attempt success rate | During placement
  First attempt vein puncture defined as single vein puncture and possibility of blood aspiration.

SECONDARY OUTCOMES:
Confirmation of tip placement in the lower 1/3 of the superior vena cava at or above the superior vena cava/right atrium junction will be performed by chest x-ray or other tip confirmation system/device and documented | During placement
  Once the PICC placement is inserted, confirmation of catheter tip location in the lower 1/3 of the superior vena cava at or above the superior vena cava/right atrium junction will be performed by chest x-ray or other tip confirmation system/device and documented. The number of adjustments to the inserted PICC needed to achieve proper tip location will be recorded
Percent of PICCs that remain in place through the required therapy time period | 90 days
  PICCs remaining in place through the required therapy time period were defined as PICCs that were either still in place at the end of the 90-day observation or had been removed because the therapy was completed (end of useful medical use), changed or cancelled.
Incidence of symptomatic venous thrombosis in patients with a PICC | 90 days
  Incidence of symptomatic venous thrombosis defined as any new occurrence of symptomatic venous thrombosis defined by thrombus presence by ultrasonography or other imaging.
Incidence of Catheter-related Bloodstream Infection | 90 days
  Incidence of Catheter-related bloodstream infection where Catheter-related bloodstream infection is defined as positive blood culture(s) with a pathogen not related to another source or positive blood culture(s) with pathogen matching catheter tip culture or blood cultures from peripheral venous puncture and PICC positive with the same pathogen.
Occurrence of complications not directly related to the cannulation procedure | 90 days
  Incidence of phlebitis where phlebitis is defined inflammation of the cannulated vessel identified by redness, swelling, warmth, tenderness, and/or cord formation.
  Incidence of extravasation where extravasation is defined as accidental infiltration of a vesicant or chemotherapeutic drug into the tissue around the catheter.
  Incidence of local infection where local infection is defined as presence of pus at the exit site and/or culture confirmed site infection.
  Incidence of accidental dislodgement where accidental dislodgement is defined as catheter accidentally dislodged the extent to which it requires replacement.
PICC lumen patency | 90 days
  Once the PICC placement is complete, the operator will confirm patency by aspirating each lumen for blood return and flushing each lumen with at least 10 mL of 0.9% NaCl.
  For inpatients, each lumen will be assessed for patency at least every 24 hours and/or before administration of medicines. Patency observations will be documented.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No